CLINICAL TRIAL: NCT02114814
Title: TRIAD-2 Center for Health Disparities Research: A Family-Based Diabetes Intervention for Hispanic Adults in an Emerging Community
Brief Title: A Family-Based Diabetes Intervention for Hispanic Adults in an Emerging Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); University of North Carolina, Greensboro (Other)
Responsible Party: Principal Investigator, Jie Hu, Principal Investigator, Ohio State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P20MD002289-06 (NIH); 2P20MD002289-06 (NIH)
Record Dates: First submitted 2014-04-03; First posted 2014-04-15 (Estimated); Results first posted 2021-02-02 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 Diabetes; Hispanic adults; Diabetes self-management; Family-based intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): Diabetes self-management and family support
  Interventions: Behavioral: Diabetes self-management program for Hispanics and their families
- Attention control group (Active Comparator): General health information
  Interventions: Behavioral: General health educational program for Hispanics and their families

INTERVENTIONS:
Behavioral: Diabetes self-management program for Hispanics and their families — The intervention group received an 8-weekly culturally tailored diabetes self-management and family support education program delivered in Spanish
  Arms: Intervention group
Behavioral: General health educational program for Hispanics and their families — The attention control group received 8-weekly education program on general health information
  Arms: Attention control group

SUMMARY:
The aim of this study was to compare the efficacy of an intervention and an attention control group in producing changes in diabetes self-management, glycemic control (HbA1c) and health related quality of life in Hispanics with type 2 diabetes.

Hypothesis: The experimental group who receive an 8 week intervention program would show significantly greater improvements than an attention control group at 1 and 6 months after the intervention in: behavioral influences of diabetes knowledge, diabetes self-efficacy, and family support, outcomes of self-reported management of diabetes (physical activity, diet, medications, and glucose monitoring), HbA1c levels, and psychological outcomes of health-related quality of life.

DETAILED DESCRIPTION:
A total of 186 participants and their family members were recruited, 103 in the experimental group and 83 in the attention control group.

An intervention consisted of eight weekly interactive modules, for a total of 12 hours, and based on modules from National Standards for Diabetes Self-Management Education, and the National Diabetes Education Program. Data were collected at baseline, immediately post-intervention, and at 3 and 6 month follow-up visits.

ELIGIBILITY:
Inclusion Criteria for participants:

1. Community-dwelling
2. Self-identification as Hispanic
3. Age 18 years or older
4. Self-identification as having a medical diagnosis of type 2 diabetes
5. An adult family member willing to participate in the study.
6. Must be able to speak either English or Spanish

Inclusion criteria for family members/relatives are:

1. Family member is over 18
2. Reside in the same household as the participant with diabetes
3. Must be able to speak either English or Spanish

Exclusion Criteria:

We will exclude Hispanic adults and family members who are:

1. diagnosed with type 1 diabetes
2. report prior (within the past year) or current participation in other diabetes self-management intervention programs
3. cognitively impaired (not oriented to time, place, or person, or with known dementia)
4. Pregnant at the time of T1 (baseline) data collection

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jie Hu, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University College of Nursing, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hu J, Amirehsani KA, Wallace DC, McCoy TP, Silva Z. A Family-Based, Culturally Tailored Diabetes Intervention for Hispanics and Their Family Members. Diabetes Educ. 2016 Jun;42(3):299-314. doi: 10.1177/0145721716636961. Epub 2016 Mar 8. PMID 26957533
- See also: A Family-Based, Culturally Tailored Diabetes Intervention for Hispanics and Their Family Members — https://www.ncbi.nlm.nih.gov/pubmed/26957533

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who had T2DM and their family members were recruited at 6 sites including clinics, physician offices, and churches in rural counties in central North Carolina between June 2012 and May 2015.
Groups:
- Intervention: A Family-Based Diabetes Self-Management Intervention
- Attention Control: General Health Education
Period: Overall Study
Arm/Group | Intervention | Attention Control
Started | 103 | 83
Completed | 88 | 74
Not Completed | 15 | 9

BASELINE CHARACTERISTICS:
Groups:
- Family-based Diabetes Intervention: The family-based intervention consisted of eight weekly group sessions for participants with diabetes and family members and two sessions (baseline and T4) with the family for data collection.
- Attention Control: Participants and their family members in the attention control group received eight weekly group sessions on general health information and two sessions with the family for data collection in addition to usual care.
- Total: Total of all reporting groups
Arm/Group | Family-based Diabetes Intervention | Attention Control | Total
Number analyzed (Participants) | 103 | 83 | 186
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 94 | 80 | 174
  >=65 years | 9 | 3 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 53 | 118
  Male | 38 | 30 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Self-reported ethnicity
  Participants
    Hispanic or Latino | 103 | 83 | 186
    Not Hispanic or Latino | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] — Body Mass Index in kg/m2
  kg/m2 | 30.9 (5.7) | 31.6 (4.6) | 31.2 (5.2)
Systolic Blood pressure [Mean (Standard Deviation); unit: mmHg] — Systolic blood pressure (SBP) was measured in mean scores in mmHg ranging from 100 mmHg to 190mmHg.
  Participants were considered hypertensive if they used antihypertensive medications or had blood pressure ≥130/80 mmHg.
  mmHg | 128.6 (18.3) | 133.1 (11.0) | 130.6 (15.6)
Physical Activity (the Short International Physical Activity Questionnaire) [Mean (Standard Deviation); unit: MET min/week] — Physical Activity (PA) was measured using the Short International Physical Activity Questionnaire (IPAQ) form, Spanish version, Last 7 Days Recall.Total physical activity metabolic equivalent of minutes/week are estimated (MET min/wk). High MET min/wk indicates high level of physical activity.
  MET min/week | 4983.1 (6906.2) | 3932.0 (5871.2) | 4514.9 (6425.5)
Dietary Intake ( BFRSS fruits/vegetables) servings/day [Mean (Standard Deviation); unit: servings/day] — Diet was assessed using questions about frequency of fruits and vegetables consumption within the Behavioral Risk Factor Surveillance Survey (BRFSS).Fruits/vegetables consumed/day were calculated with its frequencies. Total mean scores were used ranging from 0 to 5. High number refers to high fruits and vegetables consumption/day.
  servings/day | 2.6 (0.4) | 2.7 (0.4) | 2.6 (0.4)
Family Support (Supportive Resources (CIRS)) [Mean (Standard Deviation); unit: scores on a scale] — Family support was examined using the brief Chronic Illness Resources Survey (CIRS), Spanish version. The CIRS asks items on a 5-point Likert scale ranging from 1-5 that assesses social-environmental support of family members and friends, neighborhood, and community to the person with Type 2 diabetes in medication taking and exercise and diet in the past 6 months. Total mean scores were used. Higher scores indicate stronger perceived family support.
  scores on a scale | 1.4 (0.3) | 1.7 (0.4) | 1.6 (0.4)
Diabetes self-efficacy (DSE) [Mean (Standard Deviation); unit: scores on a scale] — The Stanford Diabetes Self-Efficacy (DSE), Spanish version, is an 8-item scale that measures the confidence of a person with diabetes to manage diet, exercise, and blood sugar and maintain control over the diabetes. Each of the 8 items are measured on a 10-point Likert type rating response scale ranging from 1-10. The 8 items were averaged together to calculate a total score. Higher scores indicate higher self-efficacy.
  scores on a scale | 6.4 (1.8) | 6.8 (2.4) | 6.6 (2.1)
Diabetes self-management (Revised Summary of Diabetes Self-Care Activities) [Mean (Standard Deviation); unit: days/week] — Diabetes self-management was measured by the Revised Summary of Diabetes Self-Care Activities (SDSCA), Spanish version, which assessed diet, exercise, glucose testing, medication, and foot care over the past 7 days. The mean number of days per week of diabetes self-care activities were calculated ranging from 0-7, with higher scores indicating better diabetes self-management.
  days/week
    Diabetes self-management: Diet | 3.0 (1.5) | 3.2 (1.4) | 3.1 (1.4)
    Diabetes self-management:General diet | 3.0 (1.9) | 3.3 (2.1) | 3.1 (2.0)
    Diabetes self-management: Blood glucose | 1.8 (2.3) | 1.7 (2.1) | 1.7 (2.3)
    Diabetes self-management: Foot check | 2.6 (2.4) | 4.1 (2.5) | 3.3 (2.5)
    Diabetes self-management: Medication | 6.1 (2.1) | 6.6 (1.3) | 6.3 (1.8)
Diabetes knowledge (Spoken Knowledge of Diabetes in Low Literacy Patients with Diabetes ) [Mean (Standard Deviation); unit: scores on a scale] — Diabetes knowledge was measured by the Spoken Knowledge of Diabetes in Low Literacy Patients with Diabetes (SKILLD),which assesses knowledge of glucose management, lifestyle modifications, recognition and treatment of acute complications, and activities to prevent long-term consequences of the disease.This is a verbally administered scale consisting of 10 items with scores ranging from 0 to 10 where higher scores indicate better diabetes knowledge.Total mean scores were calculated.
  scores on a scale | 2.9 (2.5) | 4.2 (2.2) | 3.5 (2.4)
Medical Outcomes Study Short Form Health Survey Version 2 (SF-12v2) [Mean (Standard Deviation); unit: scores on a scale] — Health-related quality of life was measured by the Spanish version of the Medical Outcomes Study Short Form Health Survey Version 2 (SF-12v2).29 The SF-12v2 assessed self-reported health-related quality of life through physical (PCS) and mental (MCS) component summaries. The SF-12v2 uses Likert rating scales. The PCS and MCS scores were transformed ranging from 0-100. High scores indicate better perceived health-related quality of life. Total mean scores were calculated.
  scores on a scale
    SF-12v2 PCS | 48.9 (9.2) | 47.5 (7.7) | 48.3 (8.6)
    SF-12v2 MCS | 45.9 (10.2) | 50.2 (12.7) | 47.8 (11.5)
HbA1c [Mean (Standard Deviation); unit: percent] — Glycemic control was measured with glycosylated hemoglobin A1C. Higher percent indicates worse diabetes control. The total mean scores were calculated.
  percent | 8.5 (2.1) | 9.5 (2.0) | 8.9 (2.1)

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1C
Description: Glycemic control in %.
Time Frame: Week 0 (Baseline)
Population: Hispanic adults with type 2 diabetes and their family members
Measure: Mean (95% Confidence Interval); unit: mean percentage of HbA1c
Groups:
- Intervention: Diabetes Self-Management
Arm/Group | Intervention | Attention Control
Number analyzed (Participants) | 103 | 83
mean percentage of HbA1c | 8.5 [7.9 to 9.1] | 9.4 [8.3 to 10.1]

2. Primary Outcome: Hemoglobin A1c
Description: Glycemic control
Time Frame: Month 2 (post-intervention)
Measure: Mean (95% Confidence Interval); unit: percentage of HbA1c
Arm/Group | Intervention Group | Attention Control Group
Number analyzed (Participants) | 90 | 78
percentage of HbA1c | 7.7 [7.1 to 8.2] | 8.7 [8.1 to 9.3]

3. Primary Outcome: Hemoglobin A1c
Description: Glycemic control
Time Frame: Month 3 (one month post-intervention)
Measure: Mean (95% Confidence Interval); unit: Mean percentage of HbA1c
Arm/Group | Intervention | Attention Control
Number analyzed (Participants) | 88 | 74
Mean percentage of HbA1c | 7.7 [7.1 to 8.3] | 9.0 [8.3 to 9.6]

4. Primary Outcome: Hemoglobin A1c
Description: Glycemic control
Time Frame: Month 9 (6 months post-intervention)
Measure: Mean (95% Confidence Interval); unit: Mean percentage of HbA1c
Arm/Group | Intervention | Attention Control
Number analyzed (Participants) | 82 | 67
Mean percentage of HbA1c | 8.4 [7.8 to 9.0] | 8.2 [7.7 to 8.8]

5. Secondary Outcome: Health-related Quality of Life (SF-12)
Description: The Medical Outcomes Study Short Form Health Survey Version 2 (SF-12). Physical Components Summary (PCS) and Mental Components Summary (MCS) were normed ranging from 0-100 with higher scores corresponding to better perceived health-related quality of life.
Time Frame: Week 0 (Baseline)
Measure: Mean (95% Confidence Interval); unit: Score on the PCS & MCS subscales (0=100)
Arm/Group | Intervention | Attention Control
Number analyzed (Participants) | 100 | 80
Score on the PCS & MCS subscales (0=100)
  SF-12 Physical Health (PCS) | 49.5 [47.2 to 51.8] | 49.1 [46.9 to 51.3]
  SF-12 Mental Health (MCS) | 47.2 [44.7 to 49.8] | 50.0 [46.8 to 53.3]

6. Secondary Outcome: Health-related Quality of Life (SF-12)
Description: Medical Outcomes Study Short Form Health Survey Version 2 (SF-12) Physical Components Summary (PCS) and Mental Components Summary (MCS) scores were normed ranging from 0-100 with higher scores corresponding to better perceived health-related quality of life.
Time Frame: Month 2 (post-intervention)
Measure: Mean (95% Confidence Interval); unit: Scores on PCS & MCS scores (0-100)
Arm/Group | Intervention | Attention Control
Number analyzed (Participants) | 90 | 78
Scores on PCS & MCS scores (0-100)
  SF-12 Physical Health (PCS) | 50.6 [48.8 to 52.4] | 49.5 [47.4 to 51.5]
  SF-12 Mental Health (MCS) | 47.7 [45.3 to 50.1] | 51.7 [49.1 to 54.4]

7. Secondary Outcome: Health-related Quality of Life (SF-12)
Description: as for outcome 6
Time Frame: Month 3 (one month post-intervention)
Measure: Mean (95% Confidence Interval); unit: scores on PCS & MCS scores (0-100)
Arm/Group | Intervention | Attention Control
Number analyzed (Participants) | 88 | 74
scores on PCS & MCS scores (0-100)
  SF-12 Physical Health (PCS) | 51.1 [49.4 to 52.8] | 49.6 [47.5 to 51.7]
  SF-12 Mental Health (MCS) | 47.9 [45.5 to 50.4] | 52.4 [49.8 to 55.0]

8. Secondary Outcome: Health-related Quality of Life (SF-12)
Description: The Medical Outcomes Study Short Form Health Survey, the SF-12 PCS and MCS scores were normed ranging from 0-100 with higher scores corresponding to better perceived health-related quality of life
Time Frame: Month 9 (6 months post-intervention)
Measure: Mean (95% Confidence Interval); unit: Scores on PCS & MCS scores (0-100)
Arm/Group | Intervention | Attention Control
Number analyzed (Participants) | 82 | 67
Scores on PCS & MCS scores (0-100)
  SF-12 Physical Components Summary (PCS) | 53.3 [51.4 to 55.1] | 50.3 [47.2 to 53.5]
  SF-12 Mental Components Summary (MCS) | 48.9 [45.9 to 52.0] | 55.7 [52.0 to 59.4]

ADVERSE EVENTS:
Time Frame: 9 months
Groups:
- Intervention: Family-based diabetes self-management
Arm/Group | Intervention | Attention Control
All-Cause Mortality (participants affected / at risk) | 0/103 | 0/83
Serious Adverse Events (participants affected / at risk) | 0/103 | 0/83
Other Adverse Events (participants affected / at risk) | 0/103 | 0/83

LIMITATIONS AND CAVEATS:
The study used a quasi-experimental design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No